CLINICAL TRIAL: NCT05932537
Title: Technical Description of the Ablation of Subcutaneous Contraceptive Implants in the Operating Room
Brief Title: Ablation of Subcutaneous Contraceptive Implants in the Operating Room
Acronym: TAICS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1032
Record Dates: First submitted 2022-12-14; First posted 2023-07-06 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Contraceptive Usage
Keywords: subcutaneous contraceptive implants; ablation; operating room
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subcutaneous contraceptive implants: patients who have benefited from explantation of a subcutaneous contraceptive implant in the gynecology operating room
  Interventions: Procedure: Preoperative visualization techniques

INTERVENTIONS:
Procedure: Preoperative visualization techniques — describe techniques for pre-operative visualization of subcutaneous contraceptive implants

SUMMARY:
The ablation of subcutaneous contraceptive implants is usually performed in consultation under local anesthesia. However, it happens that the implant was placed too deeply or that it migrated too deeply making it impossible to remove it in consultation. These patients should then be referred to reference centers so that the explantation takes place in the operating room. The investigators propose to describe their techniques for preoperative visualization of the implant and their techniques for surgical explantation for educational purposes.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* patient who underwent explantation of a subcutaneous contraceptive implant in the gynecology operating room
* intervention between 2018 and 2022
* person having expressed his non-opposition

Exclusion Criteria:

* explantation outside the operating room
* inability to understand the information given
* person deprived of liberty
* person under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study covers all patients who underwent explantation of a subcutaneous contraceptive implant in the gynecology operating room of the Hôpital Femme Mère Enfant, between 2018 and 2022.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound for visualization of implants | preoperatively
  Percentage of patients with an ultrasound to visualize the implants

CONTACTS AND LOCATIONS:
Locations (1):
- Gynaecology Department, Hôpital Femme Mère Enfant, Hospices Civils de Lyon, Bron, France